CLINICAL TRIAL: NCT01816945
Title: The Momba Mobile Application-based Community
Acronym: MOMBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1207010574
Record Dates: First submitted 2013-02-26; First posted 2013-03-22 (Estimated); Results first posted 2021-05-18 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-04

CONDITIONS: Mental Health Wellness 1
Keywords: Depression; Stress; Social support; Social capital; Maternal
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Access to MOMBA web-based application (Experimental): Study will provide the subject with a smartphone, pay the data plan, and facilitate access to the web-based application for purposes of researching the acceptability of the application, the operating and functioning of it, and its impact on maternal mental health.
  Interventions: Behavioral: MOMBA web-based application
- Smartphone only (No Intervention): Study will provide the subject with a smartphone and pay the data plan. Weekly assessments are completed through internet survey links sent via text message.

INTERVENTIONS:
Behavioral: MOMBA web-based application — Web-based, interactive, social network application.
  Arms: Access to MOMBA web-based application

SUMMARY:
The investigators' mobile application-based community, termed Momba, will provide a bi-directional flow of information on maternal and infant mental health to traditionally underrepresented groups of mothers and their infants. The overall goal of this mobile application-based community of low-income postpartum women and infants is to increase the social support, social networks, and social capital of low-income mothers; thereby, leading to a positive change in the health behaviors, utilization of health services, and mental health status of both mothers and their infants.

ELIGIBILITY:
Inclusion Criteria:

* Women will be recruited in their third trimester of pregnancy from Yale-New Haven Hospital (YNHH) and followed for 8 months postpartum.
* Women are eligible if they are over the age of 18, in their third trimester of pregnancy, will deliver a baby at YNHH and receive prenatal care at the Women's Center.
* Meet criteria for minor or major depressive disorder.

Exclusion Criteria:

* Mothers are not eligible to participate if they have previously given birth
* Are placing the baby for adoption
* Are planning to move in the next 18 months
* Are actively suicidal, psychotic or unable to provide informed consent

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Megan V Smith, DrPH, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
Started | 23 | 24
Completed (Completed 12 months of the intervention) | 21 | 19
Not Completed | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only | Total
Number analyzed (Participants) | 23 | 24 | 47
Age, Customized [Count of Participants; unit: Participants]
  Age category: 18-25 | 12 | 12 | 24
  Age category: 26+ | 11 | 12 | 23
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 24 | 47
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race / Ethnicity: White, Non-Hispanic | 3 | 3 | 6
  Race / Ethnicity: Black or African American, Non-Hispanic | 18 | 16 | 34
  Race / Ethnicity: White, Hispanic | 2 | 3 | 5
  Race / Ethnicity: Black or African American, Hispanic | 0 | 2 | 2
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 47
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — The Patient Health Questionnaire (PHQ-9) is 9 item questionnaire that is used to assess depression severity. The scores range from 0-27. A score of 10 or higher can be indicative of a moderate - severe level of depression severity.
  units on a scale | 7.74 (5.34) | 11.25 (6.21) | 9.53 (6.0)

OUTCOME MEASURES:

1. Primary Outcome: Phone Retention
Description: To determine the potential feasibility of providing smartphones to participants and delivering and intervention through the smartphone, phone retention was measured. Phone retention was defined as the ability of participants to retain the phone over the study period. Outcome measure used was how many participants did not need a replacement phone during the study period.
Time Frame: 15 months
Measure: Count of Participants; unit: Participants
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
Number analyzed (Participants) | 23 | 24
Participants
  Received 1 phone | 9 | 15
  Received a replacement phone | 14 | 9
Statistical Analysis 1: Comparison: Access to MOMBA Web-based Application vs Smartphone Only; Test type: Superiority; p = 0.15, Fisher Exact

2. Primary Outcome: Test the Proper Operating and Functioning of the MOMBA Application
Description: To Test the proper operating and functioning of the MOMBA application, the number of participants that received training was assessed. Intervention subjects were trained (together) on the operating and functions (including how to use the privacy settings) of the Momba application and the phone. The control subjects were trained (together) on how to complete the control questionnaires and how to use the phone.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
Number analyzed (Participants) | 23 | 24
Participants
  Number of participants trained to use phone | 23 | 24
  Number of participants who did not receive training | 0 | 0

3. Secondary Outcome: Acceptability and Performance of Structured Questionnaires
Description: To determine the acceptability and performance of structured questionnaires, the measurement is categorized into whether participants did or did not complete the 12 month follow-up interview.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
Number analyzed (Participants) | 23 | 24
Participants
  Participants who completed a 12 month follow-up interview | 20 | 19
  Participants who did not completed a 12 month follow-up interview | 3 | 5

4. Other Pre Specified Outcome: Patient Health
Description: Improve maternal emotional health, was measured by the PHQ-9. The Patient Health Questionnaire (PHQ-9) is a 9 item questionnaire that is used to assess depression severity. The scores range from 0-27. A score of 10 or higher can be indicative of a moderate - severe level of depression severity.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
Number analyzed (Participants) | 20 | 20
score on a scale | 5.6 (4.75) | 5.68 (6.37)
Statistical Analysis 1: Comparison: Access to MOMBA Web-based Application vs Smartphone Only; Two-sample t-test for PHQ-9 at 12 months; Test type: Superiority; p = 0.96, t-test, 2 sided

5. Other Pre Specified Outcome: Confident Network Score
Description: To assess the improvement maternal emotional health, the Kendler Social Support Interview was used. The Kendler Social Support Interview has scores that range from 0-5, with 5 indicating a larger social network or confidant network size. Presented below are the confident network score at 12 month follow-up.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
Number analyzed (Participants) | 20 | 20
score on a scale | 2.35 (1.39) | 1.5 (1.1)
Statistical Analysis 1: Comparison: Access to MOMBA Web-based Application vs Smartphone Only; Two-sample t-test for Social Network Score at 12 month; Test type: Superiority; p = 0.043, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Access to MOMBA Web-based Application | Smartphone Only
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes